CLINICAL TRIAL: NCT01609049
Title: Open-label, Multicenter, Non-Comparative, Prospective Observational Study to Evaluate Efficacy and Safety of Combined Ribavirin and Peginterferon Alfa-2a (40 kDa) Therapy in Patients With Chronic Hepatitis C (CHC) or Compensated Liver Cirrhosis in Real Clinical Practice
Brief Title: An Observational Study of Peginterferon Alfa-2a in Combination With Ribavirin in Participants With Chronic Hepatitis C and Compensated Liver Cirrhosis
Acronym: STANDART
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27851
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with Chronic Hepatitis C: Naive and previously treated participants who received peginterferon alfa-2a in combination with ribavirin as per local labeling requirements.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Administration of treatment will be according to local recommendation under local labeling.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin tablets twice daily orally will be administered depending on body weight, according summary product characteristics and prescribing of ribavirin in real clinical practice.
  Other Names: Copegus

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of peginterferon alfa-2a in combination with ribavirin in participants with chronic hepatitis C, including participants with compensated liver cirrhosis, in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Serologically confirmed chronic hepatitis C (CHC), hepatitis C virus (HCV) RNA detectable
* Compensated liver cirrhosis (Child-Pugh Class A) included
* Initiating combined therapy with peginterferon alfa-2a and ribavirin

Exclusion Criteria:

* Human immunodeficiency virus (HIV) co-infection
* Contraindications for combined therapy according to actual prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic hepatitis C and compensated liver cirrhosis (Class A by Child-Pugh scale) initiating treatment with Peginterferon alfa-2a and ribavirin
Sampling Method: Probability Sample
Enrollment: 1496 (Actual)
Dates: Start 2011-12-07 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) (less than [<] 50 International Units per Milliliter [IU/mL]) 24 Weeks Post Therapy Completion | Baseline up to 24 Weeks Post Therapy Completion (approximately 3.5 years)

SECONDARY OUTCOMES:
Percentage of Naive Participants With Sustained Virological Response (SVR)) and Negative HCV RNA (< 50 IU/mL) at Week 4 and 12 | Week 4, 12
Percentage of Previously Treated Participants With SVR and Negative HCV RNA (< 50 IU/mL) at Week 12 | Week 12
Percentage of Previously Treated Participants With SVR and Decrease in HCV RNA by Greater Than or Equal to (>/=) 2 Logarithm 10 From Baseline at Week 12 | Baseline, Week 12
Percentage of Naive Participants With SVR and Decrease in HCV RNA by >/= 2 Logarithm 10 From Baseline at Week 12 | Baseline, Week 12
Percentage of Previously Treated Participants With SVR, Decrease in HCV RNA by Negative HCV RNA (<50 IU/mL) at Week 24 | Week 24
Percentage of Naive Participants With SVR, Decrease in HCV RNA by Negative HCV RNA (<50 IU/mL) at Week 24 | Week 24
Percentage of Participants With SVR and Dose Reduction of Ribavirin or Peginterferon alfa-2a due to Adverse Event | Baseline up to approximately 3.5 years
Percentage of Participants With Adverse Events | Baseline up to approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (57):
- Russia (56):
  - Altay Region Aids Center, Barnaul
  - Barnaul City Hospital #5; Therapy, Barnaul
  - Chelyabinsk State Medical Academy; Infectious Diseases, Chelyabinsk
  - Chita State Medical Academy, Chita
  - Irkutsk Regional Consulting and Diagnostic Clinical Center; Regional Center of Reumatolodic Deasise, Irkutsk
  - Kaluga regional AIDS center, Kaluga
  - Kazan State Medical University, Kazan'
  - Kemerovo City Infectious Clinical Hospital; Infectious, Kemerovo
  - Khabarovsk-1 Road Clinical Hospital; Gastroenterology, Khabarovsk
  - Aids Center; Infectious, Khabarovsk
  - Kirov Region Aids-Center; Infectious, Kirov
  - Clinical Center for the Prevention and Control of AIDS and Infectious Diseases, Krasnodar
  - Specialized clinical infectious hospital, Krasnodar
  - Region Cinical Hospital; Gastroenterology, Krasnoyarsk
  - Krasnoyarsk Region Aids Center; Hepatology, Krasnoyarsk
  - Lipetsk Region Aids Center, Lipetsk
  - The scientific-research institute of epidemiology, Moscow
  - Central Medicosanitary Dept #165, Moscow
  - Russian Uni of People'S Friendship, Med. Faculty; City Clinical Hospital No 64, Internal Diseases, Moscow
  - Central Clinical Hospital of RAS ; HEPATOLOGY, Moscow
  - FGBU "Polyclinic #1 Administration President RF, Moscow
  - I.M. Sechenov First Moscow State Medical University, The V.H.Vasilenko Clinic, Moscow
  - I.M. Sechenov First Moscow State Medical University: The E.M. Tareyev Clinic, Moscow
  - Hosital of Infectious Disease #1, Moscow
  - State Medical Stomatological Uni ; Infectious, Moscow
  - Russian Medical Academy of Postgraduate Education on Botkin S.P. ; City Clinical Hospital, Moscow
  - City Hospital # 24; Hepatology, Moscow
  - Clinical hospital Centrosouz, Moscow
  - 3-D Military Clinical Hospital, Moscow
  - Medelitconsulting; Medical, Moscow
  - AIDS Center, Nizniy Novgorod
  - Infections Deseases Hospital #1, Novosibirsk
  - Baranov Republican Hospital, Petrozavodsk
  - City Hospital #1 After Semashko N.A., Rostov-on-Don
  - Rostov State Medical Uni ; Infectious Diseases, Rostov-on-Don
  - City Hospital #2; Nefrology, Rostov-on-Don
  - Ryazan State Medical University Named after I.P.Pavlov, Ryazan
  - S.P. Botkin Clinical Infectious Disease Hospital, Saint Petersburg
  - Military Medical Academy; Infectious Deseases, Saint Petersburg
  - City polyclinic №107, Saint Petersburg
  - Research institute of influenza named after I.I.Mechnikov, Saint Petersburg
  - St. Petersburg Aids Center; Haepatology, Saint Petersburg
  - Samara State Medical Uni ; Hepatogastroenterology, Samara
  - MC Gepatolog, Samara
  - City Clinical Hospital №2; Infectional diseases department, Saratov
  - Saratov Region Aids Center; Infectious Diseases, Saratov
  - Stavropol State Medical Academy, Stavropol
  - Consulting diagnostic center, Tyumen
  - State Medical Uni of Republic Bashkortostan; Infection Diseases, Ufa
  - Vladivostok state medical university, Vladivostok
  - MUZ City Clinical Infectional Hospital, Vladivostok
  - Volgograd Regional Aids Center For Aids and Infectious Diseases T Volgograd, Volgograd
  - Regional Clinical Hospital of Infectious Diseases, Voronezh
  - Yakutsk City Hospital, Yakutsk
  - Ekaterinburg Regional Hospital #1; Gastroenterology, Yekaterinburg
  - National Center for Prevention and Control of AIDS and Infectious Diseases, Yoshkar-Ola
- Dongnam Inst.of Radiological & Medical Sciences, Busan, South Korea